CLINICAL TRIAL: NCT04677725
Title: Brazilian Registry of Atherothrombotic Disease
Brief Title: NEtwork to Control ATherothrombosis (NEAT Registry)
Acronym: NEAT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital do Coracao (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: NEAT
Record Dates: First submitted 2020-12-08; First posted 2020-12-21 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Disease; Peripheral Arterial Disease; Atherothrombosis
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
NEAT is an observational cohort (Prospective registry of real world data) of patients with coronary and peripheral artery disease in an outopatient setting.

DETAILED DESCRIPTION:
National multicenter registry in Brazil with initial plan of 25 sites from the 5 Brazilian regions. It will be coordinated by HCOR Research Institute which will perform regulatory, data and site management beyond academic leadership.NEAT is an observational cohort (Prospective registry of real world data) of patients with coronary and peripheral artery disease in an outopatient setting with 12 months of follow-up with collection of data at baseline, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

Patients ≥45 years followed in ambulatory setting with ≥1 of the following 3 criteria:

1. Documented coronary disease (≥1 criteria must apply):

   * Stable angina
   * History of Unstable Angina
   * History of coronary angioplasty/stenting
   * History of coronary artery bypass graft
   * Myocardial infarction within the last 20 years
2. Documented symptomatic Peripheral Arterial Disease (≥1 criteria must apply):

   * Previous aorto-femoral bypass surgery, limb bypass surgery, or percutaneous transluminal angioplasty revascularization of the iliac, or infra-inguinal arteries, or
   * Previous limb or foot amputation for arterial vascular disease, or
   * History of intermittent claudication and one or more of the following: 1) An ankle/arm blood pressure (BP) ratio < 0.90, or 2) Significant peripheral artery stenosis (≥50%) documented by angiography, or by duplex ultrasound.

Exclusion Criteria:

* Patients from institutions that don't provide the Institutional Authorization Term,
* Incapacity of follow-up in one year according to investigator judgment (severe neuropsychiatric condition, life expectancy < 12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary and peripheral arterial disease in an outpatient setting
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients receiving evidence based therapies to reduce cardiovascular risk | Baseline
  DOMAIN 1: Appropriate use of antithrombotic therapy
Percentage of patients receiving evidence based therapies to reduce cardiovascular risk | Baseline
  DOMAIN 2: Cholesterol control
Percentage of patients receiving evidence based therapies to reduce cardiovascular risk | Baseline
  DOMAIN 3: Blood pressure control
Percentage of patients receiving evidence based therapies to reduce cardiovascular risk | Baseline
  DOMAIN 4: Glycemic control / diabetes treatment
Percentage of patients receiving evidence based therapies to reduce cardiovascular risk | Baseline
  DOMAIN 5: Weight control
Percentage of patients receiving evidence based therapies to reduce cardiovascular risk | Baseline
  DOMAIN 6: Non-pharmacological intervention: In this domain, there are 2 items to be evaluated: 1) No smoking; 2) Physical exercise ≥ 150 minutes per week.

SECONDARY OUTCOMES:
Percentage of patients receiving complete evidence based therapies to reduce cardiovascular risk | 6 and 12 months
  Patient should receive all of the following to consider complete evidence based therapy: Appropriate use of antithrombotic therapy; Cholesterol control; Blood pressure control; Glycemic control / diabetes treatment; Weight control; Non-pharmacological intervention
Percentage of patients with complete control of risk factors (blood pressure, cholesterol and glycemia) | baseline, 06 and 12 months
  blood pressure, cholesterol and glycemia levels at baseline, 06 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pedro de Barros e Silva, MD, MHS, PhD, Principal Investigator — Faculty
Locations (1):
- Hospital Do Coração, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] de Barros E Silva PGM, do Nascimento CT, Pedrosa RP, Nakazone MA, do Nascimento MU, de Araujo Melo L, Junior OLS, Zimmermann SL, de Melo RMV, Bergo RR, Precoma DB, Tramujas L, Lima EG, Dantas JMM, do Amaral Baruzzi AC, Flumignan RLG, de Oliveira Paiva MSM, Gowdak LHW, de Carvalho PN, de Figueiredo Neto JA, Silvestre OM, Fioranelli A, Vieira RD', Horak ACP, Miyada DHK, Kojima FCS, de Oliveira JS, de Oliveira Silva L, Pavanello R, Ramacciotti E, Lopes RD; NEAT Investigators. Primary results of the brazilian registry of atherothrombotic disease (NEAT). Sci Rep. 2024 Feb 20;14(1):4222. doi: 10.1038/s41598-024-54516-9. PMID 38378735